CLINICAL TRIAL: NCT06226116
Title: Comparative Study of Bone Implant Contact (BIC) With Experimental Bioecth® Surface Implant Between Native Bone and Regenerated Bone With Autogenous Dentine.
Brief Title: COMPARATIVE STUDY OF BONE IMPLANT CONTACT (BIC) ON NEW BONE REGENERATED WITH AUTOGENOUS DENTIN AND NATIVE BONE
Acronym: BIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Hernán López Sacristán, Clinical professor of master bucal surgery, implantology and periodontology, Universidad de León
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULE-034-2018
Record Dates: First submitted 2023-12-20; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Bone Resorption; Bone Regeneration
Keywords: bone implant contact; autologous dentin; socket preservation; bone density area
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- socket preservation with autologous dentin (Experimental)
  Interventions: Procedure: socket preservation; Procedure: placement of experimental implants; Procedure: histological sample collection
- extract teeth socket (Placebo Comparator): only stabilized blood clot
  Interventions: Procedure: placement of experimental implants; Procedure: histological sample collection

INTERVENTIONS:
Procedure: socket preservation — After the tooth extraction the investigator will select two sockets, one will be assigned as the experimental side and we will preserve it with cold-processed autologous dentin. The second will be designated the control group and we will only stabilize the blood clot.
  Arms: socket preservation with autologous dentin
Procedure: placement of experimental implants — After four months of preservation, titanium cylinders measuring 2 mm wide by 8 mm long, with a Bioetch® surface, will be placed.
Procedure: histological sample collection — Biopsy with trephine of a bone portion of 4mm in diameter and 10mm in length, which includes the titanium cylinder inside.
  Placement of conventional implant 5mm wide by 10mm long.

SUMMARY:
The healing process after tooth removal involves bone remodelling which implies some loss of alveolar bone volume.Among materials proposed for minimising this remodelling and preserving the bone, autologous dental tissue is a promising option, but more data are needed. In this context, the investigator evaluated size and density changes using cone beam computed tomography in autologous dental material (ADM)-preserved sockets compared to controls,and assessed biological responses by histological analysis of bone implant contact (BIC) an Area density (AA) using experimental Bioetch® surface implant.

DETAILED DESCRIPTION:
30 patients will be selected for the study, based on the inclusion/exclusion criteria and the clinical judgment of the investigator. Prior to enrollment, all subjects will be asked sign an informed consent form to demonstrate that the patient understand the scope of the study (including surgical interventions and the potential risks involved), allowing the opportunity to ask questions related to the study and giving information about treatments alternatives.

Inclusion criteria:

Partially or totally edentulous patients for whom treatment is indicated. At least 18 years of age, of both sexes and of any race. That the the participants understand that are involved in the study, including the visit requirements of follow-up.

With 6 mm or more bone width, which will be sufficient to place a cylindrical implant with 2 mm Bioetch® surface. in diameter and 8 mm of length. After 16 weeks explantation will be performed for the study, followed by placement of a wider implant.

Exclusion criteria:

Smokers. Pregnancy. History of uncontrolled systemic disease or chronic diseases. Coagulation disorder or taking anticoagulants. Treatment with bisphosphonates. Subjects with severe compromise of the immune system. History of mental instability that hinders participation in the study. Other conditions that the investigator may feel the patient is not a good candidate for this study (e.g., alcoholism, drug addiction).

Implant material: 2 mm diameter and 8 mm. of length cylinders will be used in the study. The body will be threaded with a pitch of 0.25mm. and with Bioetch® subtraction surface. The cylinders will be placed after the passage of the milling cutter. Lance and the 1.8 mm diameter. The implant enters the bed because its head It is machined with a knurled key figure that adjusts the universal screwdriver.

After 16 weeks, the study cylinders will be explanted with a trephine drill. Internal diameter 4 mm and external 4.5 mm which, in most cases, ensures recovery of the cylinder with osseointegrated material around it along its entire length.

Next, the trephine bur, with the material inside, is placed in formaldehyde buffered at 10% for transfer to the laboratory.

The patient will receive a 5 mm implant. in diameter, to rehabilitate the area where it has been collected the sample.

3 - Histological methodology: The collected sample will be placed in buffered formalin and then sent to the Histology laboratory, Anatomy section of the Department of Surgery, Medical Sciences and Social Services of the University of Alcala, for processing. This will be done in the following way:

1. Inclusion of the sample in plastic polymers of tissue section.
2. Histological preparations with undecalcified bone sections and with the implant included.
3. Cutting the samples with the EXACT system. Histological study of the sections with the description and differentiation of bone tissue in each sample.
4. Staining of the sections with toluidine blue, hematoxylin-eosin and/or trichrome.
5. Evaluation of the presence or absence of inflammatory reaction or foreign body reaction.
6. Histomorphometric study of the sample based on the morphology of the surface of the implant. The sample will be evaluated with the MIP-4 program evaluating the percentage of osseointegration (BIC), taking into account the area around the implant.
7. Statistical study to evaluate differences between the two types of samples with test analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Partially or totally edentulous patients for whom treatment is indicated
* At least 18 years of age, of both sexes and of any race.
* That they understand that they are involved in the study, including the visit requirements of follow-up.
* With 6 mm. or more bone width, which will be sufficient to place a cylindrical implant with 2 mm Bioetch® surface. in diameter and 8 mm. of length. After 16 weeks Explantation will be performed for the study, followed by placement of a wider implant.

Exclusion Criteria:

* Smokers.
* Pregnancy.
* History of uncontrolled systemic disease or chronic diseases.
* Coagulation disorder or taking anticoagulants.
* Treatment with bisphosphonates.
* Subjects with severe compromise of the immune system.
* History of mental instability that hinders participation in the study.
* Other conditions that the investigator may feel the patient is not a good candidate for this study (e.g., alcoholism, drug addiction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
BIC | 16 weeks after implant placement
  Histomorphometric study of the sample based on the morphology of the surface of the implant. The sample will be evaluated with the MIP-4 program evaluating the percentage of osseointegration (BIC), taking into account the area around the implant.
AA Bone density area | 16 weeks after implant placement
  evaluation of bone density in 0.25 mm around the experimental implant using the MIP-4 program

CONTACTS AND LOCATIONS:
Locations (1):
- centro odontológico de formación integral de León, León, Spain

IPD SHARING:
Plan to Share IPD: No